CLINICAL TRIAL: NCT00145327
Title: A 3-year, Double-blind Extension to CZOL446H2301 to Evaluate the Long-term Safety and Efficacy of Zoledronic Acid in the Treatment of Osteoporosis in Postmenopausal Women Taking Calcium and Vitamin D
Brief Title: Double-blind Extension of HORIZON Pivotal Fracture Trial (Zoledronic Acid in the Treatment of Postmenopausal Osteoporosis)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CZOL446H2301E1
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Results first posted 2011-04-20 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Osteoporosis
Keywords: Osteoporosis, Zoledronic Acid
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Zoledronic Acid 6 (Experimental): Patients who received Zoledronic acid for 3 years in the core study (CZOL446H2301; NCT00049829) received a single intravenous infusion of 5 mg Zoledronic acid once a year for 3 years (at Months 36, 48 and 60) in this extension study for a total of 6 years of treatment.
  Interventions: Drug: Zoledronic Acid
- Zoledronic Acid 3 Placebo 3 (Placebo Comparator): Patients who were treated with Zoledronic acid for 3 years in the core study received a single intravenous matching Placebo infusion once a year for 3 years in this extension study.
  Interventions: Drug: Placebo
- Placebo 3 Zoledronic Acid 3 (Experimental): Patients who were treated with placebo for 3 years in the core study received 5 mg Zoledronic acid in a single intravenous infusion once a year for 3 years (at Months 36, 48 and 60) in this extension study.
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid — Zoledronic Acid 5 mg in 100 mL physiologic 0.9% normal saline for intravenous infusion.
  Other Names: Reclast, Aclasta
  Arms: Placebo 3 Zoledronic Acid 3; Zoledronic Acid 6
Drug: Placebo — 100 mL physiologic 0.9% normal saline for intravenous infusion.
  Other Names: Reclast, Aclasta
  Arms: Zoledronic Acid 3 Placebo 3

SUMMARY:
This extension study is designed to assess the long term safety and efficacy of zoledronic acid in postmenopausal women with osteoporosis who have participated in the CZOL446H2301 (NCT00049829): HORIZON Pivotal Fracture Trial. This extension study began after the 3-year core study ended. Baseline is the same as Year 3.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received 3 infusions in the HORIZON-Pivotal Fracture (PFT) Study.

Exclusion Criteria:

* Poor kidney, eye, or liver health
* Use of certain therapies for osteoporosis in the HORIZON-PFT study (other than the study medication)
* Abnormal calcium levels in the blood

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 68 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2456 (Actual)
Dates: Start 2005-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Sponsor GmbH
Locations (31):
- United States (30):
  - Southern Arizona VA, Tucson, Arizona
  - University of Arkansas for Medical Science, Little Rock, Arkansas
  - Osteoporosis Medical Center, Beverly Hills, California
  - Osteoporosis Prevention Center, San Diego, California
  - Diablo Clinical Research, Inc, Walnut Creek, California
  - Colorado Center for Bone Research, Lakewood, Colorado
  - CRIA Research, Fort Lauderdale, Florida
  - Radiant Research, Stuart, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - United Osteoporosis Centers (UOC), Gainesville, Georgia
  - Northwestern University Center for Clinical Research, Chicago, Illinois
  - School of Medicine, Indianapolis, Indiana
  - Medical Specialist Clinical Research Center, Munster, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Maine Center for Osteoporosis Research and Education, Bangor, Maine
  - Osteoporosis Clinical Trial Center, Hagerstown, Maryland
  - Clinical Pharmacology Study Groups, Worcester, Massachusetts
  - Washington University Center for Clinical Studies, St Louis, Missouri
  - New Mexico Clinical Research and Osteoporosis Center Inc, Albuquerque, New Mexico
  - Winthrop U Hospital, Mineola, New York
  - Odyssey Research Services/CCRC Internal Medical, Fargo, North Dakota
  - University of Cincinnati Bone Health and Osteoporosis Center, Cincinnati, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Radiant Research, Wyomissing, Pennsylvania
  - Rhode Island Hospital, Endocrinology Clinical Research Unit, Providence, Rhode Island
  - University of Tennessee Health Science, Memphis, Tennessee
  - McGuire Veterans Affairs Medical Center, Richmond, Virginia
  - VA Commonwealth University, Richmond, Virginia
  - Puget Sound Osteoporosis Center, Seattle, Washington
- Novartis, Nuremberg, Germany

REFERENCES:
- [Derived] Eastell R, Boonen S, Cosman F, Reid IR, Palermo L, Cummings SR, Black DM. Relationship between pretreatment rate of bone loss and bone density response to once-yearly ZOL: HORIZON-PFT extension study. J Bone Miner Res. 2015 Mar;30(3):570-4. doi: 10.1002/jbmr.2361. PMID 25214069
- [Derived] Black DM, Reid IR, Boonen S, Bucci-Rechtweg C, Cauley JA, Cosman F, Cummings SR, Hue TF, Lippuner K, Lakatos P, Leung PC, Man Z, Martinez RL, Tan M, Ruzycky ME, Su G, Eastell R. The effect of 3 versus 6 years of zoledronic acid treatment of osteoporosis: a randomized extension to the HORIZON-Pivotal Fracture Trial (PFT). J Bone Miner Res. 2012 Feb;27(2):243-54. doi: 10.1002/jbmr.1494. PMID 22161728

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an international, multicenter, randomized, double-blind 3-year extension study in postmenopausal women with osteoporosis who had completed participation in the CZOL446H2301 (NCT00049829) core study. The extension study started 17 May 2005 (First patient enrolled) and ended 24 Nov 2009 (Last patient completed).
Pre-assignment Details: Patients who were receiving zoledronic acid in the core study were randomized in a 1:1 fashion to receive either zoledronic acid or placebo in the extension study.
  Patients who were receiving placebo in the core study were assigned to zoledronic acid in the extension study in order to retain the core study blind.
Period: Overall Study
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Started | 616 (Group Z6 and Group Z3P3 have randomized participants.) | 617 | 1223 (Group P3Z3 have non-randomized participants)
Completed | 474 | 493 | 975
Not Completed | 142 | 124 | 248
Not completed — Withdrawal by Subject | 77 | 72 | 164
Not completed — Death | 26 | 18 | 30
Not completed — Adverse Event | 14 | 11 | 22
Not completed — Lost to Follow-up | 9 | 14 | 14
Not completed — Administrative problems | 12 | 9 | 13
Not completed — Protocol Violation | 2 | 0 | 2
Not completed — Abnormal laboratory value(s) | 1 | 0 | 2
Not completed — Missing - not stated | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3 | Total
Number analyzed (Participants) | 616 | 617 | 1223 | 2456
Age Continuous [Mean (Standard Deviation); unit: Years] | 75.5 (4.88) | 75.5 (4.89) | 75.6 (4.95) | 75.5 (4.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 616 | 617 | 1223 | 2456
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Bone Mineral Density (BMD) of Femoral Neck at Year 6 Relative to Year 3
Description: The primary efficacy variable was the percentage change in BMD of the femoral neck as measured by dual x-ray absorptiometry (DXA) at Year 6 relative to Year 3. It was derived as 100 *(femoral neck BMD at Year 6 - femoral neck BMD at Year 3) / (femoral neck BMD at Year 3).
Time Frame: Year 3 (Extension Baseline; Month 36 prior to the first treatment of the extension study) and Year 6 (Month 72; end of extension study)
Population: Modified intent-to-treat (MITT) population. The MITT population included all patients in the ITT population who had DXA measurements of the femoral neck at Year 3 and Year 6. This was the primary population for primary efficacy parameter.
Measure: Mean (Standard Error); unit: Percentage Change in BMD
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Number analyzed (Participants) | 451 | 470 | 507
Percentage Change in BMD | 0.557 (0.2154) [0.43 to 1.65] | -0.493 (0.2249) [NA to NA] | 3.337 (0.2329)

2. Secondary Outcome: Bone Resorption and Formation Biochemical Markers at Year 4.5: P1NP
Description: The amount of serum n-terminal propeptide of type I collagen (P1NP) as determined by the central laboratory.
Time Frame: Year 4.5
Population: Intention to treat (ITT) population included all patients who were randomized or enrolled in the extension study at Visit 8. The number of patients analyzed = the number of patients with measurements at Year 4.5 as determined by the analysis window.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Number analyzed (Participants) | 433 | 460 | 870
ng/mL | 18.842 (0.4325) [0.59 to 0.65] | 29.677 (0.6977) [NA to NA] | 17.256 (0.3743)

3. Secondary Outcome: Bone Resorption and Formation Biochemical Markers at Year 6: P1NP
Description: The amount of serum P1NP as determined by the central laboratory
Time Frame: Year 6
Population: Intention to treat (ITT) population included all patients who were randomized or enrolled in the extension study at Visit 8. The Number of patients analyzed = the number of patients with measurements in Year 6 as determined by the analysis window.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Number analyzed (Participants) | 392 | 414 | 426
ng/mL | 27.356 (0.6340) | 30.344 (0.6050) | 25.926 (0.7765)

4. Secondary Outcome: Percentage Change in BMD of Lumbar Spine at Year 4.5 Relative to Year 3
Description: The percentage change in BMD as measured by DXA at Year 4.5 relative to Year 3. It was derived as 100 * (BMD at Year 4.5 - BMD at Year 3)/(BMD at Year 3).
Time Frame: Year 3 (Extension Baseline; Month 36 prior to the first treatment of the extension study) and Year 4.5 (Month 54)
Population: Intention to treat (ITT) population included all patients who were randomized or enrolled in the extension study at Visit 8. The number of patients analyzed = the number of patients with measurements at Year 4.5 and Year 3 as determined by the analysis window.
Measure: Mean (Standard Error); unit: Percentage Change in BMD
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Number analyzed (Participants) | 101 | 102 | 195
Percentage Change in BMD | 2.618 (0.384) [0.38 to 2.42] | 1.196 (0.3510) [NA to NA] | 6.551 (0.3035)

5. Secondary Outcome: Percentage Change in BMD of Lumbar Spine at Year 6 Relative to Year 3
Description: The percentage change in BMD as measured by DXA at Year 6 relative to Year 3. It was derived as 100 * (BMD at Year 6 - BMD at Year 3)/(BMD at Year 3).
Time Frame: Year 3 (Extension Baseline; Month 36 prior to the first treatment of the extension study) and Year 6
Population: Intention to treat (ITT) population included all patients who were randomized or enrolled in the extension study at Visit 8. The number of patients analyzed = the number of patients with measurements at Year 6 and Year 3 as determined by the analysis window.
Measure: Mean (Standard Error); unit: Percentage change in BMD
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Number analyzed (Participants) | 100 | 84 | 128
Percentage change in BMD | 3.473 (0.4653) | 1.606 (0.4550) | 8.875 (0.5398)

6. Secondary Outcome: Percentage Change in BMD of Distal Radius at Year 4.5 Relative to Year 3
Description: as for outcome 4
Time Frame: Year 3 (Extension Baseline; Month 36 prior to the first treatment of the extension study) and Year 4.5 (Month 54)
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Percentage change in BMD
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Number analyzed (Participants) | 100 | 99 | 188
Percentage change in BMD | 0.378 (0.3615) | -0.924 (0.3158) | 0.386 (0.3071)

7. Secondary Outcome: Percentage Change in BMD of Distal Radius at Year 6 Relative to Year 3
Description: as for outcome 5
Time Frame: Year 3 (Extension Baseline; Month 36 prior to the first treatment of the extension study) and Year 6 (Month 72)
Population: as for outcome 5
Measure: Mean (Standard Error); unit: Percentage change in BMD
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Number analyzed (Participants) | 96 | 82 | 125
Percentage change in BMD | 0.178 (0.3661) | -0.567 (0.4025) | 0.299 (0.3473)

8. Secondary Outcome: Percentage Change in BMD of Femoral Neck, Total Hip and Trochanter at Year 4.5 Relative to Year 3
Description: The percentage change in BMD as measured by DXA at 4.5 relative to Year 3. It was derived as 100 * (BMD at Year 4.5 - BMD at Year 3)/(BMD at Year 3).
Time Frame: Year 3 (Extension Baseline; Month 36 prior to the first treatment of the extension study) and Year 4.5 (Month 54)
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Percentage change in BMD
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Number analyzed (Participants) | 525 | 544 | 1047
Percentage change in BMD
  Femoral Neck | 0.738 (0.1874) | 0.210 (0.2058) | 2.697 (0.1516)
  Total Hip | 0.479 (0.1337) | -0.070 (0.1354) | 3.228 (0.1244)
  Trochanter | 0.813 (0.1919) | 0.041 (0.1936) | 4.611 (0.2050)

9. Secondary Outcome: Percentage Change in BMD of Femoral Neck, Total Hip and Trochanter at Year 6 Relative to Year 3
Description: as for outcome 5
Time Frame: Year 3 (Extension Baseline; Month 36 prior to the first treatment of the extension study) and Year 6 (Month 72)
Population: as for outcome 5
Measure: Mean (Standard Error); unit: Percentage change in BMD
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Number analyzed (Participants) | 451 | 470 | 570
Percentage change in BMD
  Femoral Neck | 0.577 (0.2154) [0.58 to 2.15] | -0.493 (0.2249) [NA to NA] | 3.337 (0.2329)
  Total Hip | 0.083 (0.1647) [0.80 to 2.14] | -1.151 (0.1817) [NA to NA] | 3.815 (0.1877)
  Trochanter | 0.628 (0.2275) [1.56 to 3.44] | -0.903 (0.2462) [NA to NA] | 6.072 (0.2894)

10. Secondary Outcome: Percentage of Patients With New and New/Worsening Morphometric Vertebral Fractures
Description: Lateral vertebral x-rays were performed at the final core study visit and at Year 6 and read by a central expert reader at a central imaging laboratory to assess for new or new/worsening morphometric vertebral fracture. The percentage of patients with new morphometric vertebral fractures (observed for the first time) and patients with either new or worsening morphometric vertebral fractures was calculated.
Time Frame: Year 3 (Extension Baseline; Month 36 prior to the first treatment of the extension study) and Year 6
Population: Intention to treat (ITT) population included all patients who were randomized or enrolled in the extension study at Visit 8. The number of patients analyzed = the number of patients with measurements at Year 6 as determined by the analysis window.
Measure: Number; unit: Percentage of patients
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Number analyzed (Participants) | 469 | 486 | 585
Percentage of patients
  New morphometric vertebral fracture | 3.0 [0.26 to 0.90] | 6.2 [NA to NA] | 2.9
  New/Worsening morphometric vertebral fracture | 3.4 | 7.0 | 3.1

11. Secondary Outcome: Number of Participants With Incidence of Clinical Fracture
Description: Clinical fracture excludes finger, toe, and facial bone fractures. Clinical vertebral fracture includes thoracic spine fracture and lumbar spine fracture. Non-vertebral fracture excludes clinical vertebral, finger, toe, and facial bone fractures.
Time Frame: Extension Baseline (Year 3; Month 36) to Year 6
Population: Intention to treat (ITT) population included all patients who were randomized or enrolled in the extension study at Visit 8. n = the number of patients with measurements at Year 6 as determined by the analysis window.
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Number analyzed (Participants) | 616 | 617 | 1223
Participants
  Clinical fracture | 51 (8.15) | 51 (8.52) | 91
  Clinical vertebral fractures | 7 | 4 | 7
  Non-vertebral fractures | 45 | 47 | 85
  Hip fracture | 7 | 8 | 10

12. Secondary Outcome: Qualitative Bone Biopsy Parameters
Description: Unpaired transiliac crest bone biopsy was performed for histomorphometry, which was obtained after double tetracycline labeling. No data were collected for Patients who received Placebo for the first 3 years of the study (Placebo 3 Zoledronic Acid 3).
Time Frame: End of Study Visit at Year 6
Population: Bone Biopsy sub-population.
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Number analyzed (Participants) | 3 | 2 | 0
Participants
  Osteomalacia | 0 | 0 |
  Woven bone | 0 | 0 |
  Cortical trabeculation | 0 | 0 |
  Marrow fibrosis | 0 | 0 |
  Normal mineralization and normal osteoid | 3 | 2 |
  Contained double labeling | 3 | 2 |

13. Secondary Outcome: Change in Serum Creatinine From Baseline to 9-11 Days Post Year 3 Infusion
Description: Serum creatinine measurements performed by a central laboratory was used to evaluate acute changes in renal function 9-11 days after study drug infusion in Z6 patients compared to Z3P3 patients and in P3Z3 patients.
Time Frame: Extension Baseline (Year 3; Month 36 prior to the first treatment of the extension study) to 9-11 days after the Year 3 infusion
Population: Safety Population included all patients in the ITT population who received at least one dose of study drug during the extension study.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Number analyzed (Participants) | 613 | 616 | 1221
μmol/L | 1.96 (9.364) | 1.28 (8.757) | 0.21 (12.360)

14. Secondary Outcome: Change in Serum Creatinine From Baseline to 9-11 Days Post Year 4 Infusion
Description: Serum creatinine measurements performed by a central laboratory was used to evaluate acute changes in renal function 9-11 days after Year 4 study drug infusion.
Time Frame: Extension Baseline (Year 3; Month 36 prior to the first treatment of the extension study) to 9-11 days after the Year 4 infusion
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Number analyzed (Participants) | 613 | 616 | 1221
μmol/L | 3.35 (23.580) | 2.23 (9.891) | 2.47 (13.042)

15. Secondary Outcome: Change in Serum Creatinine From Baseline to 9-11 Days Post Year 5 Infusion
Description: Serum creatinine measurements performed by a central laboratory was used to evaluate acute changes in renal function 9-11 days after Year 5 study drug infusion.
Time Frame: Extension Baseline (Year 3; Month 36 prior to the first treatment of the extension study) to 9-11 days after the Year 5 infusion
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Number analyzed (Participants) | 613 | 616 | 1221
μmol/L | 3.46 (21.735) | 0.71 (10.278) | 1.04 (11.882)

16. Secondary Outcome: The Number of Participants With Clinically Significant Laboratory Parameters
Description: Evaluate the laboratory key profile such as Calcium, Creatinine and Urea. The number of patients with clinically significant calcium, creatinine and urea were reported.
Time Frame: Extension Baseline (Year 3; Month 36 prior to the first treatment of the extension study) to Year 6
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Number analyzed (Participants) | 612 | 615 | 1210
Participants
  Creatinine <18 μmol/L | 1 | 0 | 1
  Creatinine >221 μmol/L | 3 | 0 | 2
  Calcium <1.87 mmol/L | 0 | 0 | 1
  Calcium >2.89 mmol/L | 4 | 0 | 4
  Urea < 0.7 mmol/L | 0 | 0 | 0
  Urea >14.3 mmol/L | 9 | 10 | 17

ADVERSE EVENTS:
Time Frame: Extension Baseline (Year 3; Month 36) to Year 6
Description: Adverse events and serious adverse events were based on the safety population which includes all patients in the ITT population who received at least one dose of study drug during the extension study.
Arm/Group | Zoledronic Acid 6 | Zoledronic Acid 3 Placebo 3 | Placebo 3 Zoledronic Acid 3
Serious Adverse Events (participants affected / at risk) | 191/613 | 168/616 | 297/1221
Other Adverse Events (participants affected / at risk) | 421/613 | 427/616 | 908/1221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 6 (N=613) | Zoledronic Acid 3 Placebo 3 (N=616) | Placebo 3 Zoledronic Acid 3 (N=1221)
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 5
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 4
Angina pectoris (Cardiac disorders) | 3 | 1 | 6
Angina unstable (Cardiac disorders) | 0 | 2 | 1
Aortic valve disease (Cardiac disorders) | 0 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 12 | 7 | 10
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 1
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 2 | 0 | 4
Bundle branch block left (Cardiac disorders) | 0 | 0 | 2
Cardiac arrest (Cardiac disorders) | 2 | 2 | 2
Cardiac disorder (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 4 | 1 | 9
Cardiac failure congestive (Cardiac disorders) | 3 | 2 | 5
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 3 | 2 | 4
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 2
Myocardial fibrosis (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 5 | 4 | 5
Myocardial ischaemia (Cardiac disorders) | 2 | 0 | 2
Palpitations (Cardiac disorders) | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 2 | 3
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 2
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 0 | 1
Deafness bilateral (Ear and labyrinth disorders) | 0 | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 1
Ototoxicity (Ear and labyrinth disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 3 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0
Goitre (Endocrine disorders) | 1 | 1 | 0
Thyrotoxic crisis (Endocrine disorders) | 0 | 1 | 0
Amaurosis fugax (Eye disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 4 | 6 | 13
Eye disorder (Eye disorders) | 0 | 0 | 1
Eye inflammation (Eye disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 1 | 0 | 0
Hyalosis asteroid (Eye disorders) | 0 | 1 | 0
Retinal artery embolism (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 2
Sympathetic ophthalmia (Eye disorders) | 0 | 1 | 0
Trichiasis (Eye disorders) | 1 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 8
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 0 | 1
Anal polyp (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1 | 5
Colonic stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 4
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 3
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Femoral hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 3 | 1 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophagitis (Gastrointestinal disorders) | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 2
Hiatus hernia (Gastrointestinal disorders) | 0 | 2 | 0
Ileal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 2 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 2 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 3 | 2
Intestinal polyp (Gastrointestinal disorders) | 2 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 2 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatic duct dilatation (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0
Volvulus of small bowel (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1 | 3
Accidental death (General disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 3
Chest pain (General disorders) | 1 | 1 | 3
Chills (General disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 3
Fatigue (General disorders) | 1 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 1 | 0 | 1
Impaired healing (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 2
Multi-organ failure (General disorders) | 1 | 0 | 0
Necrosis (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 5
Oedema peripheral (General disorders) | 1 | 1 | 0
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 2
Sudden death (General disorders) | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 3 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 3 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 4 | 6 | 3
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 2
Abdominal abscess (Infections and infestations) | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 2
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 5 | 1
Bronchitis bacterial (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 3 | 2 | 1
Clostridial infection (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 5
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 1
Endometritis (Infections and infestations) | 0 | 1 | 0
Endophthalmitis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 2 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 1
Influenza (Infections and infestations) | 0 | 1 | 1
Intervertebral discitis (Infections and infestations) | 0 | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 2 | 0 | 0
Osteomyelitis chronic (Infections and infestations) | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 10 | 5 | 13
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 0
Post procedural pneumonia (Infections and infestations) | 0 | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 2 | 3
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 2
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 2
Device breakage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Device dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 2 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 4 | 7
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 3 | 2 | 5
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 2 | 0
Fractured ischium (Injury, poisoning and procedural complications) | 2 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 1 | 2 | 2
Hip fracture (Injury, poisoning and procedural complications) | 5 | 7 | 5
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 3 | 5
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 2 | 2
Mouth injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 5 | 5 | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pubic rami fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 5
Rib fracture (Injury, poisoning and procedural complications) | 2 | 1 | 4
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 5 | 0 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 4 | 4
Barium enema (Investigations) | 0 | 0 | 1
Blood glucose decreased (Investigations) | 1 | 0 | 0
Blood osmolarity decreased (Investigations) | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 3
International normalised ratio decreased (Investigations) | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 2
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Lipomatosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4 | 3
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 4 | 13
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4 | 1
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 2 | 6
Carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 3
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to chest wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Morton's neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mucoepidermoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Urinary bladder adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1
Anoxic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0
Basal ganglia infarction (Nervous system disorders) | 0 | 0 | 1
Brain injury (Nervous system disorders) | 1 | 0 | 0
Brain stem haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebral artery embolism (Nervous system disorders) | 0 | 1 | 0
Cerebral artery occlusion (Nervous system disorders) | 0 | 0 | 2
Cerebral haemorrhage (Nervous system disorders) | 2 | 0 | 2
Cerebral infarction (Nervous system disorders) | 0 | 2 | 4
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0
Cerebrosclerosis (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 6 | 3 | 8
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 2 | 0 | 0
Dementia (Nervous system disorders) | 1 | 0 | 2
Diabetic coma (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 4 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 0 | 1
Encephalitis (Nervous system disorders) | 0 | 0 | 1
Encephalomyelitis (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 2 | 0 | 0
Hemiplegia (Nervous system disorders) | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 2
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 2 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Monoparesis (Nervous system disorders) | 0 | 1 | 0
Myelopathy (Nervous system disorders) | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 1 | 0 | 0
Nerve root compression (Nervous system disorders) | 0 | 0 | 1
Neurodegenerative disorder (Nervous system disorders) | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 2
Parkinsonism (Nervous system disorders) | 0 | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 1
Progressive bulbar palsy (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0
Spinal claudication (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 5
Temporal lobe epilepsy (Nervous system disorders) | 0 | 1 | 0
Thalamic infarction (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 7 | 2 | 3
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 1
Vascular dementia (Nervous system disorders) | 0 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Anxiety disorder due to a general medical condition (Psychiatric disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 2 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1
Glomerulonephritis chronic (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Bartholin's cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Breast fibrosis (Reproductive system and breast disorders) | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 1
Genital prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 1
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Rectocele (Reproductive system and breast disorders) | 1 | 1 | 0
Urogenital prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 2
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 2
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 3
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary artery stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 5
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Acrodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Immobile (Social circumstances) | 0 | 1 | 0
Social problem (Social circumstances) | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 2 | 1 | 0
Arterial disorder (Vascular disorders) | 1 | 0 | 0
Arterial stenosis limb (Vascular disorders) | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 3
Deep vein thrombosis (Vascular disorders) | 3 | 1 | 2
Embolism (Vascular disorders) | 1 | 0 | 0
Femoral arterial stenosis (Vascular disorders) | 1 | 0 | 1
Femoral artery occlusion (Vascular disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 2 | 1 | 4
Hypertensive crisis (Vascular disorders) | 2 | 2 | 3
Hypotension (Vascular disorders) | 1 | 0 | 5
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0
Shock (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1 | 1
Thrombosis (Vascular disorders) | 0 | 1 | 2
Varicose vein (Vascular disorders) | 2 | 1 | 1
Vasculitis (Vascular disorders) | 0 | 0 | 1
Vasoconstriction (Vascular disorders) | 0 | 0 | 1
Venous insufficiency (Vascular disorders) | 0 | 1 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 6 (N=613) | Zoledronic Acid 3 Placebo 3 (N=616) | Placebo 3 Zoledronic Acid 3 (N=1221)
Cataract (Eye disorders) | 35 | 43 | 72
Diarrhoea (Gastrointestinal disorders) | 31 | 32 | 57
Nausea (Gastrointestinal disorders) | 20 | 26 | 94
Fatigue (General disorders) | 24 | 20 | 64
Pyrexia (General disorders) | 30 | 19 | 181
Bronchitis (Infections and infestations) | 48 | 49 | 80
Influenza (Infections and infestations) | 32 | 31 | 63
Nasopharyngitis (Infections and infestations) | 61 | 61 | 95
Urinary tract infection (Infections and infestations) | 77 | 94 | 143
Fall (Injury, poisoning and procedural complications) | 50 | 60 | 110
Arthralgia (Musculoskeletal and connective tissue disorders) | 119 | 106 | 253
Back pain (Musculoskeletal and connective tissue disorders) | 113 | 111 | 206
Bone pain (Musculoskeletal and connective tissue disorders) | 30 | 16 | 88
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 34 | 31 | 76
Myalgia (Musculoskeletal and connective tissue disorders) | 28 | 25 | 147
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 55 | 49 | 87
Pain in extremity (Musculoskeletal and connective tissue disorders) | 51 | 54 | 121
Dizziness (Nervous system disorders) | 26 | 31 | 69
Headache (Nervous system disorders) | 37 | 40 | 125
Hypertension (Vascular disorders) | 46 | 92 | 136

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.